CLINICAL TRIAL: NCT05498220
Title: A Phase II Trial Evaluating the Efficacy of Polatuzumab Vedotin With Rituximab, Gemcitabine, Dexamethasone, and Cisplatin (PV-RGDP) Chemotherapy for Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Polatuzumab Vedotin With R-GDP in Relapsed/Refractory Diffuse Large B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2033
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Relapsed; refractory; polatuzumab vedotin; rituximab; gemcitabine; cisplatin
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — polatuzumab vedotin; Rituximab; Hyaluronoglucosaminidase; Gemcitabine; Cisplatin; Dexamethasone

STUDY DESIGN:
Intervention Model Description: The study will use a Simon two-stage design. In the first stage 27 evaluable subjects will be recruited. If there are at least 13 (≥ 13) subjects with a partial or complete response after 4 cycles, another 17 subjects will be enrolled and treated in the second stage of the trial, for a total of 44 evaluable subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): The subjects with diffuse large B-cell lymphoma were relapsed or refractory after the first treatment and receiving the study protocol treatment.
  Interventions: Drug: Polatuzumab vedotin (PV); Drug: Rituximab; Drug: Hyaluronidase; Drug: Gemcitabine; Drug: Cisplatin; Drug: Dexamethasone; Drug: GCSF

INTERVENTIONS:
Drug: Polatuzumab vedotin (PV) — 1.8 mg/kg, intravenous, at day 1, in every 21 days
Drug: Rituximab — 375 mg/m2 intravenous, at day 1 or day 2, in every 21 days
Drug: Hyaluronidase — 1,400 mg/23,400 units sub-cutaneous, starts at cycle 2, in every 21 days
Drug: Gemcitabine — 1,000 mg/m2 intravenous at day 1 and 8, in every 21 days
Drug: Cisplatin — 75 mg/m2, intravenous, at day 1, in every 21 days
Drug: Dexamethasone — 40 mg intravenous at day 1, Per oral days at days 2-4
Drug: GCSF — granulocyte-colony stimulating factor (GCSF )

SUMMARY:
This study aimed to evaluate the efficacy of a novel regimen consisting of polatuzumab vedotin in combination with rituximab, gemcitabine, dexamethasone, and cisplatin (PV-RGDP) for the treatment of diffuse large B-cell lymphoma that either came back or did not improve after the treatments (rrDLBCL).

This combination has not been approved by the Food and Drug Administration (FDA) for the treatment of rrDLBCL. Salvage therapy (treatment after standard treatment failed) needs to be improved. Rituximab, gemcitabine, dexamethasone, and cisplatin combination is a standard therapy for rrDLBCL and polatuzumab vedotin (PV) is a novel antibody-drug conjugate targeting CD79b. PV has shown efficacy in the setting of rrDLBCL and can improve the response rates of standard salvage therapy.

This study will focus on subjects in the first relapse (one prior regimen) and will include both subjects who are transplant eligible and those who are transplant ineligible.

ELIGIBILITY:
In order to participate in this study, a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria:

1. Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
2. Biopsy proven diffuse large B-cell lymphoma (DLBCL) in the first relapse (biopsy can be from initial diagnosis). The study will allow high-grade B cell lymphoma, but not including Burkitt's lymphoma.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
4. Radiologic evidence of active disease within 28 days of starting trial therapy.
5. Only one prior line of therapy.
6. Prior cancer treatment must be completed at least 14 days prior to the start of treatment and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤ Grade 1 or start of treatment.
7. Subjects may be eligible or ineligible for autologous stem cell transplant

Exclusion Criteria:

1. Known severe, active bacterial, viral, fungal, mycobacterial, parasitic, or other infections at study enrollment that may put the subject at undue risk as determined by the investigator.
2. Subjective hearing loss interfering with daily activities or evidence of greater than mild hearing loss compared to age appropriate normal on screening audiometry are excluded.
3. Women who are pregnant or breastfeeding or who intend to become pregnant within a year of the last dose of study treatment.
4. Subjects with a history of prior or concurrent second primary malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the study drugs are eligible for enrollment in the trial.
5. Previous exposure to polatuzumab vedotin.
6. History of severe allergic or anaphylactic reaction to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine.
7. Contraindication to gemcitabine or cisplatin, or dexamethasone or similar corticosteroid.
8. Symptomatic cardiac disease including ventricular dysfunction, left ventricular ejection fraction < 40%, symptomatic coronary artery disease or symptomatic arrhythmias.
9. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation > 91% on room air.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2026-11-07 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 4 months (End of Treatment)
  ORR is defined as the proportion of subjects who received the study treatment, and achieved complete response (CR) or partial response (PR) by Lugano classification.
  Complete Response: Complete metabolic response on Positron emission tomography (PET) image or Target nodes/nodal masses must regress to ≤ 1.5 cm in the largest transverse diameter (LDi) or no extra lymphatic sites of disease on Computerized Tomography (CT).
  Partial Response: Score of 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size on PET and ≥50% decrease in the sum of the products of diameters (SPD) of up to 6 target measurable nodes and extranodal sites on CT.

SECONDARY OUTCOMES:
Complete response rate (CR) | Up to 4 months (End of Treatment)
  CR is defined as the proportion of subjects who received the study treatment, achieved complete response (CR) by the Lugano classification.
Progression free survival (PFS) | Up to 2 years
  PFS is defined as the time from the start of study treatment until progression by Lugano classification or death.
  Progressive Disease: Score 4 or 5 with an increase in the intensity of uptake from baseline and/or new fluorodeoxyglucose (FDG) -avid foci consistent with lymphoma at the interim or end-of-treatment assessment on PET, or an individual node/lesion must be abnormal with LDi > 1.5 cm, increase by ≥ 50% from the cross product of the shortest axis perpendicular to LDi (SDi) nadir and an increase in LDi or SDi from nadir: 0.5 cm for lesions ≤ 2 cm, 1.0 cm for lesions > 2 cm.
Overall Survival (OS) | Up to 2 years
  OS is defined as the time from the start of treatment until death from any cause.
Number of participants with adverse events | Up to 2 years
  The number of participants with adverse events will be listed and tabulated by grade to determine the safety and toxicity.
  Adverse Events will be graded according to The National Cancer Institute (NCI) of Common Terminology Criteria for Adverse Events (CTCAE) version 5. The scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dittus, DO, MPH, Principal Investigator — Division of Hematology | Lymphoma Program Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials